CLINICAL TRIAL: NCT05609708
Title: Technological Development and Clinical Parallel Testing of Preimplantation Genetic Testing for Generalization
Brief Title: Technological Development and Clinical Parallel Testing of PGT-G
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-245-02
Record Dates: First submitted 2022-11-03; First posted 2022-11-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Genetic Disease
Keywords: PGT; stLFR-WGS
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and waste WGA products from embryos
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preimplantation genetic testing (PGT) has three different testings according to the type of genetic disease, which was classified as PGT-M, PGT-SR and PGT-A. If the couple is tested for two different genetic diseases at the same time, it is necessary to customize the probe and adopt different detection methods, which increases the cost and cycle of testing. Advanced expert pre-experimental analysis is required for PGT-M in couples with monogenic disease. If the family members are unavailable, only the polar bodies, sperms or affected embryos can be used to analysis, which not only increases the risk of failure, but also increases the difficulty of detection. At present, BGI has developed a new single-tube complete Long fragment whole genome sequencing (stLFR-WGS) technology, which uses the same molecular tag on the short read sequencing fragments from the same long DNA molecule to achieve accurate short read sequencing to obtain long DNA information. Multiple genetic abnormalities such as gene variation, chromosome aneuploidy and chromosome structure rearrangement can be directly detected in embryos without pre-experiment of family members, so as to achieve universal normalization of the three PGT methods and solve the PGT detection needs of patients with multiple genetic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing PGT cycle;
2. Patients with balanced chromosomal structural rearrangement (reciprocal translocation, Robertsonian translocation, inversion, etc.) by conventional karyotype analysis;
3. Clearly diagnosed monogenic genetic disease, and the related genes and their mutations are judged to be pathogenic or likely pathogenic;
4. Chromosomal abnormalities in recurrent abortion tissues or in PGT-A embryos; The number of blastocysts was >= 1, and the morphological classification was more than 4BC/4CB.

Exclusion Criteria:

1. Belonged to any contraindications of PGT;
2. Failed to embryo biopsy;
3. Failed to embryo WGA failure or abnormal quality control;
4. Failed to embryo sequencing, and the result was unknown.

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients with genetic diseases undergoing PGT cycle
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis specificity | 1 day (the time of sequencing)
  specificity
diagnosis sensitivity | 1 day (the time of sequencing)
  sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong Provicne, China

IPD SHARING:
Plan to Share IPD: No